CLINICAL TRIAL: NCT00852631
Title: Open-label Multicentre Study on Efficacy and Safety of Oral Quetiapine (Seroquel XR) in Adults With Schizophrenia
Brief Title: Seroquel XR in Adults With Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely terminated due to insufficient recruitment.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00060
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia
Keywords: Quetiapine efficacy in schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine fumarate (Seroquel) — 600mg Extended release tablet, oral, once daily
  Other Names: Seroquel XR

SUMMARY:
The purpose of this study is to evaluate the efficacy of Seroquel XR in schizophrenia patients with acute worsening symptoms. Consequently, to assess whether the study drug is safe and acceptable on the daily dose basis, orally given, up to 600 mg once a day for 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the DSM-IV criteria for schizophrenia
* Patient has a PANSS total score ≥ 70 at baseline
* Patient has a CGI-S score of ≥ 4(moderately ill) at baseline
* Patient is healthy on the basis of physical examination and vital signs at baseline

Exclusion Criteria:

* Positive urine drug screen for Opiates, amphetamine, barbiturate, cocaine, cannabis, or ecstasy abuse
* Has history of neuroleptic malignant syndrome, seropositive for anti-HIV, hepatitis B or C virus antigen
* Patient with unstable or inadequately treated Diabetes Mellitus
* Use of potent cytochrome P450 inhibitors or inducer within 14 days before baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thawatchai Leelahanaj, MD, Principal Investigator — Phramongkutklao Hospital, Bangkok, Thailand
Locations (3):
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Songkhla

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients provide informed consent and are screened for eligibility (at Visit 1) up to 7 days before baseline assessment on Day 1.
Pre-assignment Details: On Day 1, baseline assessments will be performed, and patients will be assigned to Seroquel XR at 300 mg. On Day 2 all patients are assigned to reach target dose of Seroquel XR at 600 mg. Administration of study medication continue with Seroquel XR 600 mg daily until Day 42. Each visit will have ± 3 days window period.
Groups:
- Seroquel XR: Seroquel XR 300mg on day 1, 600mg from day 2 onwards. The treatment period will take 6 weeks or 42 days.
Period: Overall Study
Arm/Group | Seroquel XR
Started | 28
Completed | 17
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Seroquel XR
Number analyzed (Participants) | 28
Age Continuous [Median (Standard Deviation); unit: Years] | 43 (39.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20

OUTCOME MEASURES:

1. Secondary Outcome: Change in Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: Clinical Global Impression - Severity of Illness. Maximum possible value is 7 (worst outcome), the minimum is 1 (best outcome). Values are considered better outcome: decrease from baseline > 1 score.
Time Frame: From Day 1 (Baseline) to Day 42
Population: The number of patient at Day 42 (n= 17) is different than at Baseline (n= 28), because some of them withdraw/terminate during the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 28
Scores on a scale
  Day 1 (Baseline) (n= 28) | 4.6 (0.7)
  Day 42 (n= 17) | 2.7 (1.1)

2. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Change in Positive and Negative Syndrome Scale Total Score from Day 1 (baseline) to Day 42 (final visit) or withdrawal. Minimum value of total PANSS is 30 , Maximum is 210.
  Minimum value considered better is score decreased from baseline at least 30%.
Time Frame: From Day 1 (baseline) to Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 28
Scores on a scale
  Day 1 (Baseline) (n= 28) | 85.3 (28.8)
  Day 42 (n= 17) | 48.5 (28.6)

3. Secondary Outcome: Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: as for outcome 1
Time Frame: Day 14
Population: The number of patient is different, because some of them withdraw/terminate during the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Seroquel XR
Number analyzed (Participants) | 21
Scores on a scale | 3.2 (1.1)

ADVERSE EVENTS:
Arm/Group | Seroquel XR
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel XR (N=28)
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel XR (N=28)
Dry Mouth (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Hypotension (Vascular disorders) | 3
Stiff nose (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No